CLINICAL TRIAL: NCT05615402
Title: Improving Bone Health in Wheelchair Users by a Long-term Intervention Combining Bone-specific Exercise and Nutrition
Brief Title: Intervention on Bone Health in Wheelchair Users
Acronym: BoneWheel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Sunnaas Rehabilitation Hospital (Other); Norwegian University of Science and Technology (Other); HAN University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Kristin L. Jonvik, Principal investigator, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NorwegianSSS BoneWheel
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Bone Loss; Spinal Cord Injuries; Cerebral Palsy; Spina Bifida; Dysmelia; Amputation
MeSH Terms: conditions — Bone Diseases, Metabolic; Spinal Cord Injuries; Cerebral Palsy; Spinal Dysraphism

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial over 24-weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Group A: strength training 3x/week + nutrition optimalisation
  Interventions: Other: Bone-specific strength training; Dietary Supplement: Nutrition optimalisation
- Nutrition group (Experimental): Group B: nutrition optimalisation
  Interventions: Dietary Supplement: Nutrition optimalisation

INTERVENTIONS:
Other: Bone-specific strength training — Muscular strength and rate of force development (RFD) will be assessed in the key exercises of the intervention protocol
  Arms: Training group
Dietary Supplement: Nutrition optimalisation — Dietary supplement of protein, vitamin D and Calcium 3x/w Dietary counselling based on individual dietary records

SUMMARY:
The low mechanical loading of bones among wheelchair users leads to an increased risk of bone fractures and associated complications due to low bone mineral density (BMD). Adding mechanical loading through physical activity in combination with optimizing nutrition may counteract these negative consequences in wheelchair users and thereby provide positive impact for bone health, as well as for physical and mental health.

In this project, a multidisciplinary team will tailor a bone-specific exercise and nutrition program to increase BMD in sport active and non-active wheelchair users with initial low BMD.

DETAILED DESCRIPTION:
The primary aim of this project is to investigate the effects of combined exercise training with high mechanical loading of bones and nutritional counselling for improving bone health in wheelchair users with an initially low-normal to low BMD (Z-score ≤ 0.0). Specifically, the following objectives are to determine the effects of the intervention on:

1. Bone health, measured as changes in BMD and blood bone markers.
2. Physical health, including body composition and muscular fitness.
3. Mental health, with focus on well-being, QOL and user experience.

The secondary aim is to use this knowledge to develop recommendations and implementation plans for exercise and nutrition to promote bone health of wheelchair users.

Using a randomized controlled design, participants will undergo an exercise intervention in which the participants also will receive nutritional optimization for bone remodelling. Main outcomes are change in BMD, blood bone markers, physical health and mental health parameters. Based on the outcomes of the RCT, the researchers will develop evidence-based practical health promoting recommendations and an implementation plan for health practitioners working with wheelchair users in the municipalities.

ELIGIBILITY:
Inclusion Criteria:

* BMD Z-score of the spine ≤ 0 SD
* primary aid for mobility being a manual wheelchair, i.e. ≥50% of the time
* 18-60 Y
* congenital (i.e., CP, spina bifida, dysmelia, hip dysplasia) and acquired disabilities (i.e., SCI, amputation)
* non-progressive impairment, and in the case of SCI; ≥ 2 years since time of injury
* ability to perform key exercises (e.g., overhead press)

Exclusion Criteria:

* injury acquired <2 Y ago
* change in health and/or medication within the last 3 months
* fractures affecting measured sites or contraindicating strength testing/training
* menopausal, pregnancy or planned pregnancy during the study period
* language or cognitive barriers affecting the ability to understand all aspects of the study
* • patients with progressive neurological disease, serious or uncontrollable epilepsy, endocrine diseases (including diabetes mellitus type 1 or 2, thyroid disorders, calcium homeostasis disorders and metabolic bone disease, pituitary gland disorder, sex hormone disorders), cancer, serious mental disorder, or comorbid medical conditions affecting either a) nutritional function: i.e., malabsorption problems due to previous surgery in the gastrointestinal tract, inflammatory bowel disease, coeliac disease, eating disorders, chronic pancreatitis, liver or kidney disease (those that cannot convert vitamin D to its active form in the body), other conditions affecting vitamin D or calcium absorption; b) musculoskeletal system: i.e., congenital systemic skeletal dysplasia affecting bone density, inflammatory arthritis conditions (such as rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, and lupus), ongoing tendinitis or muscle injuries not compatible with the exercise intervention; c) cardiovascular system: i.e. congenital heart failure, congenital connective tissue disorders affecting the aorta and/or arteries, other cardiovascular conditions not compatible with the exercise intervention;
* the use of certain medications: bisphosphonates, PTH (teriparatide), Denosumab, Raloksiphen, Prednisolone/steroids/androgenic steroids, high dose oestrogen (including medroxyprogesterone acetate contraceptives) immunosuppressive medications/ chemotherapies, vitamin K, anti-epileptic medication (Lamotrigine, Phenytoin, Phenobarbital, Carbamazepine, Primidone), proton pump inhibitors (PPIs), selective serotonin receptor inhibitors (SSRIs), thiazolidinediones (TZDs), anticonvulsants, hormone deprivation therapy, calcineurin inhibitors, and isotretinoin.
* other therapies that aim to increase bone mineral density, e.g., vibration therapy, functional electrical stimulation (FES)
* alternative medicine that interfere with vitamin D or calcium metabolism or affect bone mineral density
* known other contraindication of resistance exercise.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density of the spine | 24-weeks
  Z-score for L1-4

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No